CLINICAL TRIAL: NCT07302360
Title: Guselkumab Real-world Effectiveness Among Bio-NaÏve Patients With Moderate-to-severe Ulcerative Colitis in China: A Multicenter, Non-interventional, Prospective Study
Brief Title: A Real-World Study of Guselkumab in Chinese Participants With Ulcerative Colitis
Acronym: GENIUS
Status: Recruiting | Type: Observational
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CNTO1959UCO4003
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Guselkumab: Moderate to Severe Ulcerative Colitis (UC): Participants with confirmed diagnosis of moderate-to-severe UC treated with guselkumab as per standard clinical practice will be enrolled. No drug will be provided as part of this study. Only data available from standard clinical practice and medical records will be collected and observed.

SUMMARY:
The purpose of this study is to assess the measurable changes in health, function, or quality of life (clinical outcomes) after receiving guselkumab in real-world clinical practice amongst Chinese participants with ulcerative colitis (UC; a long-term disease of the large intestine in which the lining of the colon [part of large intestine] becomes inflamed and develops tiny open ulcers), who have not received biologic therapy (a medicine made from living organisms or their components) previously.

ELIGIBILITY:
Inclusion criteria:

* Has a confirmed diagnosis of moderately to severely active UC, defined as: a) baseline modified Mayo score of 4 to 9; b) screening endoscopy with Mayo endoscopic subscore (MES) greater than or equal to (>=) 2; c) Mayo rectal bleeding subscore (RBS) >= 1 at baseline
* Eligible for advanced treatment and initiate guselkumab therapy per participating physician decision in accordance with product package insert
* Have no prior exposure to advanced therapies (bio-naive), such as tumor necrosis factor (TNF)-alpha antagonists, anti-integrin agents, anti-interleukin (IL) agents, sphingosine-1-phosphate receptor modulators, janus kinase (JAK) inhibitors or their corresponding generics and biosimilars, per participating physician assessment
* Participant (and/or their legally-acceptable representative where applicable) must sign an informed consent form (ICF) allowing source data verification in accordance with local requirements

Exclusion criteria:

* Acute severe UC or infectious colitis or other conditions when patients is likely to require a colectomy
* Contraindicated to guselkumab per the label
* Currently enrolled in or plan to participate in any other clinical trials from signing informed consent to the final dose administration of guselkumab
* Participants who will be receiving guselkumab therapy combined with a second advanced therapy
* Participants with a history of colectomy and/or pouch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible Chinese participants with moderate-to-severe UC who are bio-naive will be consecutively enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Response at Week 12 | At Week 12
  Clinical response is defined as a decrease from baseline in the partial Mayo score by >= 30 percent (%) and >= 2 points, with either a >=1 decrease from baseline in rectal bleeding subscore (RBS) or an RBS of 0 or 1. Partial Mayo score is a non-invasive clinical measure for determining the severity of UC. The total score falls between 0 and 9, where higher score indicates more severity.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Response at Week 24 and Week 48 | At Week 24 and Week 48
  Clinical response is defined as a decrease from baseline in the partial Mayo score by >= 30 % and >= 2 points, with either a >=1 decrease from baseline in RBS or an RBS of 0 or 1. Partial Mayo score is a non-invasive clinical measure for determining the severity of UC. The total score falls between 0 and 9, where higher score indicates more severity.
Percentage of Participants Achieving Symptomatic Response at Week 2 | At Week 2
  Symptomatic response is defined as a decrease from induction baseline in the patient reported outcome (PRO)-2 by at least 30% and at least 1 point, with either at least 1-point decrease from induction baseline in RBS or an RBS of 0 or 1. PRO-2 consists of the two components (rectal bleeding and stool frequency). The stool frequency subscale is rated as follows: 0 (normal stool frequency), 1 (1-2 stools more than normal), 2 (3-4 stools more than normal), and 3 (5 or more stools more than normal). The rectal bleeding subscale is rated as: 0 (no blood), 1 (streaks of blood less than half the time), 2 (obvious blood most of the time), and 3 (blood alone). Higher score indicates more severity in symptoms.
Mean Change from Baseline in Stool Frequency Subscore (SFS) Over Week 2 | From Baseline to Week 2
  SFS is a component of PRO-2. The stool frequency subscale is rated as follows: 0 (normal stool frequency), 1 (1-2 stools more than normal), 2 (3-4 stools more than normal), and 3 (5 or more stools more than normal). Higher score indicates more severity in symptoms.
Mean Change from Baseline in RBS Over Week 2 | From Baseline to Week 2
  RBS is a component of PRO-2. The rectal bleeding subscale is rated as: 0 (no blood), 1 (streaks of blood less than half the time), 2 (obvious blood most of the time), and 3 (blood alone). Higher score indicates more severity in symptoms.
Percentage of Participants Achieving Clinical Remission at Week 12, Week 24 and Week 48 | At Week 12, Week 24 and Week 48
  Clinical remission is defined as a partial Mayo score less than or equal to (<=) 2 with no sub-score greater than (>) 1. Partial Mayo score is a non-invasive clinical measure for determining the severity of UC. The total score falls between 0 and 9, where higher score indicates more severity.
Percentage of Participants Achieving Symptomatic Remission at Week 2 | At Week 2
  Symptomatic remission as measured by PRO-2 is defined as a SFS of 0 or 1 and an RBS of 0, where the SFS has not increased from induction baseline. The SFS is rated as follows: 0 (normal stool frequency), 1 (1-2 stools more than normal), 2 (3-4 stools more than normal), and 3 (5 or more stools more than normal). The RBS is rated as: 0 (no blood), 1 (streaks of blood less than half the time), 2 (obvious blood most of the time), and 3 (blood alone). Higher score indicates more severity in symptoms.
Percentage of Participants Achieving Steroid-Free Remission at Week 12, 24 and 48 | At Weeks 12, 24 and 48
  Steroid-free remission is defined as clinical remission with no use of corticosteroids for at least 30 days. Clinical remission is defined as partial Mayo score <= 2 with no sub-score >1.
Percentage of Participants Achieving Sustained Remission at Week 24 and Week 48 | At Week 24 and Week 48
  Sustained remission is defined as clinical remission maintenance status at post-induction (Week 12) in participants who had attained clinical remission by the end of the 12-week induction therapy.
Percentage of Participants with Endoscopic Improvement (Healing) at Week 24 and Week 48 | At Week 24 and Week 48
  Endoscopic improvement (healing) is defined as endoscopic remission Mayo endoscopic subscore (MES) of 0 or 1. The MES consists of 3 subscores: stool frequency, rectal bleeding and physician's global assessment, each subscore is graded from 0 (normal) to 3 (severe) with higher scores indicate more severe disease.
Percentage of Participants Achieving Endoscopic Remission (Normalization) at Week 24 and Week 48 | At Week 24 and Week 48
  Endoscopic remission (normalization) is defined as an MES of 0. The MES consists of 3 subscores: stool frequency, rectal bleeding and physician's global assessment, each subscore is graded from 0 (normal) to 3 (severe) where higher scores indicate more severe disease.
Percentage of Participants Discontinuing from Treatment | Up to Week 48
  Treatment discontinuation is defined as discontinuation of guselkumab treatment for any reason.
Percentage of Participants Switching from Treatment | Up to Week 48
  Treatment switch is defined as initiation of another medication for UC treatment after guselkumab discontinuation.
Time to Treatment Discontinuation | Up to Week 48
  Time to treatment discontinuation is defined as the time from the guselkumab start date to the time of treatment discontinuation.
Time to Treatment Switch | Up to Week 48
  Time to treatment switch is defined as the time from the guselkumab start date to the time of initiation of a new treatment other than guselkumab.
Percentage of Participants on Guselkumab Dosing Schedules of 200 Milligrams (mg) Once Every 4 Weeks (q4w) or 100 mg Once Every 8 Weeks (q8w) | From Baseline through Week 12 to Week 48
  The percentage of participants on guselkumab dosing schedules of 200mg q4w or 100 mg q8w will be assessed. For each dosing schedule, the percentage will be calculated by dividing the number of participants receiving the specific dosing regimen by the number of participants still being followed up at those time points, multiplied by 100%.
Percentage of Participants Undergoing Dose Escalation/ De-Escalation | Week 12 up to Week 48
  Percentage of participants having dose escalation/ de-escalation during maintenance treatment will be assessed. The percentage will be calculated by dividing the number of participants having dosage adjustment (that is, dose escalation/de-escalation) after Week 0 at any visit time point compared to his/her previous recorded administration dosage, multiplied by 100%.
Percentage of Participants Achieving Inflammatory Bowel Disease Questionnaire (IBDQ) Remission | At Week 12, Week 24 and Week 48
  IBDQ remission is defined as total IBDQ score >= 170. The IBDQ is a validated, 32-item, self-reported questionnaire for patients with inflammatory bowel disease that will be used to evaluate the disease-specific health-related quality of life (QoL) across 4 dimensional scores: bowel symptoms (loose stools, abdominal pain), systemic functions (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Scores range from 32 to 224, with higher scores indicating better outcomes.
Change from Baseline in C-Reactive Protein (CRP) Levels | Baseline, Week 12, Week 24 and Week 48
  Change in CRP levels since guselkumab initiation will be reported.
Change from Baseline of Fecal Calprotectin Levels | Baseline, Week 12, Week 24 and Week 48
  Change in fecal calprotectin levels since guselkumab initiation will be reported.
Percentage of Participants Achieving CRP Normalization | At Week 12, Week 24 and Week 48
  Normalization of CRP is defined as reduction of less than or equal to 5 microgram per liter (mg/L) at weeks 12, 24 and 48 since baseline. Percentage of participants with abnormal CRP at baseline achieving CRP normalization will be reported.
Percentage of Participants Achieving Fecal Calprotectin (FCP) Normalization | At Week 12, Week 24 and Week 48
  Normalization of fecal calprotectin is defined as reduction of <= 250 microgram per gram (mcg/g) at weeks 12, 24 and 48 since baseline. Percentage of participants with abnormal FCP at baseline achieving fecal calprotectin normalization will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, China

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency